CLINICAL TRIAL: NCT02672878
Title: Prospective Study of Bioresorbable Vascular Scaffold Treatment in Patients With In-stent Restenosis
Brief Title: Restenosis Intrastent: Bioresorbable Vascular Scaffolds Treatment (RIBS VI)
Acronym: RIBS VI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Spanish Society of Cardiology (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Instituto de Investigación Sanitaria Hospital Universitario de la Princesa (Other); Abbott Medical Devices (Industry); Terumo Medical Corporation (Industry)
Responsible Party: Principal Investigator, Fernando Alfonso, MD, Spanish Society of Cardiology
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RIBS VI
Record Dates: First submitted 2016-01-05; First posted 2016-02-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Coronary In-stent Restenosis
Keywords: In-stent restenosis; Bioresorbable vascular scaffold; Stent; Drug-eluting stent; Coronary angiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- BVS implantation in patients with ISR (Experimental)
  Interventions: Device: Bioresorbable vascular scaffold

INTERVENTIONS:
Device: Bioresorbable vascular scaffold

SUMMARY:
Treatment of patients with in-stent restenosis (ISR) remains a challenge. This study will assess the efficacy of Bioresorbable Vascular Scaffolds (BVS) (Abbott Vascular) in the treatment of patients suffering from ISR.

DETAILED DESCRIPTION:
Treatment of patients with ISR remains a challenge. Currently both drug-eluting stents (DES) and drug-coated balloons (DCB) are considered as the strategies of choice in this setting. However, data on the value of BVS in patients with ISR is scarce. BVS are very effective to inhibit neointimal proliferation and they avoid the need of implanting a new permanent metal layer. Accordingly, currently, there is a major interest to elucidate the potential value of BVS in patients with ISR.

This prospective Spanish multicenter study will assess the clinical and angiographic outcome of patients with ISR treated with BVS. BVS will be implanted in selected patients (fulfilling inclusion and exclusion criteria) presenting with either BMS-ISR or DES-ISR. Care will be paid to ensure device optimization. Angiographic follow-up will be obtained at 6-9 months. A centralized angiographic corelab will be used to provide QCA measurements. Clinical follow-up will be also obtained at 1 year and then yearly. Clinical events will be adjudicated by an independent Clinical Event Committee.

ELIGIBILITY:
In-stent restenosis with ischemia. Signed Informed Consent IRB approval

INCLUSION CRITERIA:

PATIENT

* Age > 20 and < 85 years of age
* Acceptance of late angiographic evaluation
* Angina or objective evidence of ischemia

LESION

* ISR (>50% diameter stenosis on visual assessment)
* Previous stent location known

EXCLUSION CRITERIA:

PATIENT

* Inclusion in other clinical research protocol
* Allergy to antiplatelet agents
* Women in childbearing age
* Severe associated systemic diseases (including renal or liver failure) or diseases affecting life expectancy
* Recent myocardial infarction
* Time from index stent implantation < 1 month
* Anticipated difficulties for late angiographic evaluation

LESION

* Stent thrombosis or large thrombus within the stent
* Angiographic failure during initial stent implantation or persistence or large dissection.
* Severe tortuosity or calcification or major difficulties during previous stent implantation
* Vessel diameter < 2.25 mm (visual assessment)
* Stenosis outside stent stent edge (edge ISR are eligible)
* Very diffuse ISR (>30 mm in length)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Minimal lumen diameter as assessed by quantitative coronary angiography at late angiographic follow-up | angiographic follow-up at 6-9 months
  This is a single arm study and results will be analyzed per arm. However, the angiographic and clinical results will be also compared with those obtained in other arms of previous RIBS trials
Combined clinical end-point (cardiac death, myocardial infarction and target vessel revascularization) | 1 year of clinical follow-up
  This is a well-accepted outcome measure of individual clinical end-points. Definition of myocardial infarction is similar to that used in previous RIBS studies.

SECONDARY OUTCOMES:
Acute gain | procedure
  Change in the minimal lumen diameter from baseline to the final procedural angiogram. Acute angiographic parameter.
Minimal lumen diameter | procedure
  Acute angiographic parameter
Percent diameter stenosis | procedure
  Acute angiographic parameter
Restenosis rate | 6-9 months
  Late angiographic parameter
Percent diameter stenosis | 6-9 months
  Late angiographic parameter
Late loss | 6-9 months
  Change in minimal lumen diameter from the final procedure to the follow-up angiogram at 6-9 months. Late angiographic parameter.
Net gain | 6-9 months
  Is the difference between acute gain and late loss. Late angiographic parameter.
Loss index | 6-9 months
  Late angiographic parameter
Combined clinical outcome measure (Cardiac death, Myocardial infarction, target lesion revascularization) | 1 year, 2 years, 3 years, 4 years, 5 years
  This is a well-accepted outcome measure of individual clinical end-points. Definition of myocardial infarction is similar to that used in previous RIBS studies.
Cardiac death | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Total mortality | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Myocardial infarction | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Target vessel revascularization | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Target lesion revascularization | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Stent thrombosis | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome
Major bleeding | 1 year, 2 years, 3 years, 4 years, 5 years
  Individual clinical outcome

CONTACTS AND LOCATIONS:
Locations (19):
- Spain (19):
  - Complexo Universitario Hospitalario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Infanta Cristina, Badajoz, Badajoz
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Complejo Asistencial de León, León, León
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Complejo Hospitalario de Toledo, Toledo, Toledo
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Hospital de Galdakao, Vizcaya, Vizcaya

REFERENCES:
- [Result] Alfonso F, Zueco J, Cequier A, Mantilla R, Bethencourt A, Lopez-Minguez JR, Angel J, Auge JM, Gomez-Recio M, Moris C, Seabra-Gomes R, Perez-Vizcayno MJ, Macaya C; Restenosis Intra-stent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. A randomized comparison of repeat stenting with balloon angioplasty in patients with in-stent restenosis. J Am Coll Cardiol. 2003 Sep 3;42(5):796-805. doi: 10.1016/s0735-1097(03)00852-0. PMID 12957423
- [Result] Alfonso F, Melgares R, Mainar V, Lezaun R, Vazquez N, Tascon J, Pomar F, Cequier A, Angel J, Perez-Vizcayno MJ, Sabate M, Banuelos C, Fernandez C, Garcia JM; Restensois Intra-stent: Ballon angioplasty versus elective Stenting (RIBS) Investigators. Therapeutic implications of in-stent restenosis located at the stent edge. Insights from the restenosis intra-stent balloon angioplasty versus elective stenting (RIBS) randomized trial. Eur Heart J. 2004 Oct;25(20):1829-35. doi: 10.1016/j.ehj.2004.07.019. PMID 15474698
- [Result] Alfonso F, Auge JM, Zueco J, Bethencourt A, Lopez-Minguez JR, Hernandez JM, Bullones JA, Calvo I, Esplugas E, Perez-Vizcayno MJ, Moreno R, Fernandez C, Hernandez R, Gama-Ribeiro V; RIBS Investigators. Long-term results (three to five years) of the Restenosis Intrastent: Balloon angioplasty versus elective Stenting (RIBS) randomized study. J Am Coll Cardiol. 2005 Sep 6;46(5):756-60. doi: 10.1016/j.jacc.2005.05.050. PMID 16139121
- [Result] Alfonso F, Perez-Vizcayno MJ, Gomez-Recio M, Insa L, Calvo I, Hernandez JM, Bullones JA, Hernandez R, Escaned J, Macaya C, Gama-Ribeiro V, Leitao-Marques A; Restenosis Intrastent: Balloon Angioplasty Versus Elective Stenting (RIBS) Investigators. Implications of the "watermelon seeding" phenomenon during coronary interventions for in-stent restenosis. Catheter Cardiovasc Interv. 2005 Dec;66(4):521-7. doi: 10.1002/ccd.20524. PMID 16261546
- [Result] Alfonso F, Cequier A, Angel J, Marti V, Zueco J, Bethencourt A, Mantilla R, Lopez-Minguez JR, Gomez-Recio M, Moris C, Perez-Vizcayno MJ, Fernandez C, Macaya C, Seabra-Gomes R; Restenosis Intra-stent Balloon angioplasty versus elective Stenting (RIBS) Investigators. Value of the American College of Cardiology/American Heart Association angiographic classification of coronary lesion morphology in patients with in-stent restenosis. Insights from the Restenosis Intra-stent Balloon angioplasty versus elective Stenting (RIBS) randomized trial. Am Heart J. 2006 Mar;151(3):681.e1-681.e9. doi: 10.1016/j.ahj.2005.10.014. PMID 16504631
- [Result] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Bethencourt A, Marti V, Lopez-Minguez JR, Angel J, Mantilla R, Moris C, Cequier A, Sabate M, Escaned J, Moreno R, Banuelos C, Suarez A, Macaya C; RIBS-II Investigators. A randomized comparison of sirolimus-eluting stent with balloon angioplasty in patients with in-stent restenosis: results of the Restenosis Intrastent: Balloon Angioplasty Versus Elective Sirolimus-Eluting Stenting (RIBS-II) trial. J Am Coll Cardiol. 2006 Jun 6;47(11):2152-60. doi: 10.1016/j.jacc.2005.10.078. PMID 16750678
- [Result] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Fernandez C, Escaned J, Banuelos C, Bethencourt A, Lopez-Minguez JR, Angel J, Cequier A, Sabate M, Moris C, Zueco J, Seabra-Gomes R; Restenosis Intra-Stent: Balloon Angioplasty Versus Elective Stent Implantation (RIBS-I) and Restenosis Intra-Stent: Balloon Angioplasty Versus Elective Sirolimus-Eluting Stenting (RIBS-II) Investigators. Sirolimus-eluting stents versus bare-metal stents in patients with in-stent restenosis: results of a pooled analysis of two randomized studies. Catheter Cardiovasc Interv. 2008 Oct 1;72(4):459-67. doi: 10.1002/ccd.21694. PMID 18814274
- [Result] Alfonso F, Perez-Vizcayno MJ, Hernandez R, Bethencourt A, Marti V, Lopez-Minguez JR, Angel J, Iniguez A, Moris C, Cequier A, Sabate M, Escaned J, Jimenez-Quevedo P, Banuelos C, Suarez A, Macaya C; RIBS-II Investigators. Long-term clinical benefit of sirolimus-eluting stents in patients with in-stent restenosis results of the RIBS-II (Restenosis Intra-stent: Balloon angioplasty vs. elective sirolimus-eluting Stenting) study. J Am Coll Cardiol. 2008 Nov 11;52(20):1621-7. doi: 10.1016/j.jacc.2008.08.025. PMID 18992651
- [Result] Alfonso F, Perez-Vizcayno MJ, Dutary J, Zueco J, Cequier A, Garcia-Touchard A, Marti V, Lozano I, Angel J, Hernandez JM, Lopez-Minguez JR, Melgares R, Moreno R, Seidelberger B, Fernandez C, Hernandez R; RIBS-III Study Investigators (under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology). Implantation of a drug-eluting stent with a different drug (switch strategy) in patients with drug-eluting stent restenosis. Results from a prospective multicenter study (RIBS III [Restenosis Intra-Stent: Balloon Angioplasty Versus Drug-Eluting Stent]). JACC Cardiovasc Interv. 2012 Jul;5(7):728-37. doi: 10.1016/j.jcin.2012.03.017. PMID 22814777
- [Result] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia Del Blanco B, Seidelberger B, Iniguez A, Gomez-Recio M, Masotti M, Velazquez MT, Sanchis J, Garcia-Touchard A, Zueco J, Bethencourt A, Melgares R, Cequier A, Dominguez A, Mainar V, Lopez-Minguez JR, Moreu J, Marti V, Moreno R, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS V Study Investigators, under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology. A randomized comparison of drug-eluting balloon versus everolimus-eluting stent in patients with bare-metal stent-in-stent restenosis: the RIBS V Clinical Trial (Restenosis Intra-stent of Bare Metal Stents: paclitaxel-eluting balloon vs. everolimus-eluting stent). J Am Coll Cardiol. 2014 Apr 15;63(14):1378-86. doi: 10.1016/j.jacc.2013.12.006. Epub 2014 Jan 8. PMID 24412457
- [Result] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia Del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Rivero F, Masotti M, Zueco J, Cequier A, Moris C, Fernandez-Ortiz A, Escaned J, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; Restenosis Intra-stent: drug-eluting Balloon vs. everolimus-eluting Stent (RIBS IV) Study Investigators (under the auspices of the Working Group on Interventional Cardiology of the Spanish Society of Cardiology). Rationale and design of the RIBS IV randomised clinical trial (drug-eluting balloons versus everolimus-eluting stents for patients with drug-eluting stent restenosis). EuroIntervention. 2015 Jul;11(3):336-42. doi: 10.4244/EIJY14M09_07. PMID 25244700
- [Result] Alfonso F, Perez-Vizcayno MJ, Cardenas A, Garcia del Blanco B, Garcia-Touchard A, Lopez-Minguez JR, Benedicto A, Masotti M, Zueco J, Iniguez A, Velazquez M, Moreno R, Mainar V, Dominguez A, Pomar F, Melgares R, Rivero F, Jimenez-Quevedo P, Gonzalo N, Fernandez C, Macaya C; RIBS IV Study Investigators (under auspices of Interventional Cardiology Working Group of Spanish Society of Cardiology). A Prospective Randomized Trial of Drug-Eluting Balloons Versus Everolimus-Eluting Stents in Patients With In-Stent Restenosis of Drug-Eluting Stents: The RIBS IV Randomized Clinical Trial. J Am Coll Cardiol. 2015 Jul 7;66(1):23-33. doi: 10.1016/j.jacc.2015.04.063. PMID 26139054
- [Derived] Alfonso F, Cuesta J, Garcia Del Blanco B, Bosa F, Perez de Prado A, Masotti M, Trillo R, Rumoroso JR, Moreno R, Cequier A, Gutierrez H, Garcia Touchard A, Lopez-Minguez JR, Zueco J, Serra A, Velazquez M, Moris C, Bastante T, Garcia-Guimaraes M, Rivero F, Fernandez-Perez C; Restenosis Intrastent: Bioresorbable Vascular Scaffolds Treatment with Scoring Balloon Pre-dilatation (RIBS VI 'Scoring') Study Investigators (under the auspices of the Interventional Cardiology Working Group of the Spanish Society of Cardiology). Scoring balloon predilation before bioresorbable vascular scaffold implantation in patients with in-stent restenosis: the RIBS VI 'scoring' study. Coron Artery Dis. 2021 Mar 1;32(2):96-104. doi: 10.1097/MCA.0000000000000904. PMID 32558692
- [Derived] Alfonso F, Cuesta J, Perez-Vizcayno MJ, Garcia Del Blanco B, Rumoroso JR, Bosa F, Perez de Prado A, Masotti M, Moreno R, Cequier A, Gutierrez H, Garcia Touchard A, Lopez-Minguez JR, Zueco J, Marti V, Velazquez M, Moris C, Bastante T, Garcia-Guimaraes M, Rivero F, Fernandez C; Interventional Cardiology Working Group of the Spanish Society of Cardiology. Bioresorbable Vascular Scaffolds for Patients With In-Stent Restenosis: The RIBS VI Study. JACC Cardiovasc Interv. 2017 Sep 25;10(18):1841-1851. doi: 10.1016/j.jcin.2017.06.064. Epub 2017 Aug 30. PMID 28866036